CLINICAL TRIAL: NCT01980433
Title: Study of Writing Improvement in Patients With Wilson Disease and Dystonia After One Session of Inhibitory Repetitive Transcranial Magnetic Stimulation
Brief Title: Inhibitory rTMS in Dystonic Wilson Patients
Acronym: WILSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P121105
Record Dates: First submitted 2013-10-24; First posted 2013-11-11 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Wilson Disease; Movement Disorders; Repetitive Transcranial Magnetic Stimulation
Keywords: Wilson disease; Dystonia; Movement Disorders; Handwriting; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Hepatolenticular Degeneration; Movement Disorders; Dystonia | interventions — Transcranial Magnetic Stimulation; Lead

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Experimental): Repetitive Transcranial Magnetic stimulation: 1 Hz rTMS, delivered to left somatosensory cortex during rest. Intervention is delivered during 20 minutes in one single session.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Other: pre and post-rTMS electroencephalogram; Other: WCRS; Other: handwriting scale DPRE; Other: visual analog scale of discomfort writing and parameters collected on touchpad
- Sham rTMS (Sham Comparator): Placebo Transcranial Magnetic stimulation delivered to left somatosensory cortex during rest. Intervention is delivered during 20 minutes in one single session.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Other: pre and post-rTMS electroencephalogram; Other: WCRS; Other: handwriting scale DPRE; Other: visual analog scale of discomfort writing and parameters collected on touchpad

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Inhibitory 1 Hz rTMS, delivered to left somatosensory cortex during rest. Intervention is delivered during 20 minutes in one single session.
Other: pre and post-rTMS electroencephalogram — to verify the absence of infraclinical seizures
Other: WCRS — Writer's cramp rating scale
Other: handwriting scale DPRE — handwriting in development and being evaluated by the NRC Wilson
Other: visual analog scale of discomfort writing and parameters collected on touchpad

SUMMARY:
Wilson disease is a genetic disorder resulting in copper accumulation in liver, brain and eye. The neurologic complications include dystonic syndrome, which is a prolonged and excessive muscle activation responsible for abnormal postures. Hand dystonia prevents daily life activities such as writing, which is particularly disabling, since writing is the only mean of communication in these patients with significant slurred speech. Treatment is limited and only partially effective.

Low frequency (<or=1Hz) repetitive transcranial magnetic stimulation (rTMS) has shown inhibiting properties when applied over the cortex. Since dystonia has been correlated to hyperactivation of the neurons of the somatosensory cortex (SSC), we hypothesize that one single 20-minute session of 1 Hz rTMS applied on left SSC will improve writing of the right dystonic hand, assessed immediately at the end of the session.

DETAILED DESCRIPTION:
This study investigates the handwriting performance of an homogeneous cohort of patients with Wilson disease and right handed dystonia, after one single inhibitory repetitive transcranial magnetic stimulation (rTMS). Fifteen patients with focal right hand dystonia will receive randomly either active or sham rTMS (1 Hz) to the left somatosensory cortex (SSC) in one single 20 minutes session. Handwriting performance will be measured immediately after this unique session (Visual analogic scale of subjective discomfort in writing, DPRE and WCRS scales, pen pressure and pen velocity measured on touchpad), compared to scores obtained 24 hours before the session. Three days later, the patient will receive the other session (sham rTMS or active rTMS) and the same parameters will be evaluated.

This is a single-center, randomized, crossover, prospective, clinical and double-blind study (the rTMS session is performed by the neurophysiologist, but the patient and the neurologist who will perform the handwriting evaluation are blind to the session).

ELIGIBILITY:
Inclusion Criteria:

* Wilson disease with focal right hand dystonia
* No modification of medical treatment for 6 months
* No botulinum toxin administration within the past four months
* Right handed
* Focal right hand dystonia
* Cerebral Magnetic Resonance performed the last 6 months with no other lesion than met in Wilson disease
* Over 18
* Insurance policy holder
* Informed consent

Exclusion Criteria:

* Pregnant woman
* Guardianship procedure
* Seizure history
* Other cerebral lesions on cerebral MRI than met in Wilson Disease
* Unable to stay quiet for 30 minutes
* Handwriting impossible
* Contra-indications to repetitive Transcranial Magnetic Stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
immediate and significant improvement in writing | up to 1 week
  Improvement of handwriting performance immediately after one single 20 minutes session of inhibitory (1 Hz) repetitive transcranial magnetic stimulation over the left somatosensory cortex.
  quantitative test score of writing WCRS
  Active or sham stimulation will be randomly assigned to the patient and the other session will be performed 3 days later.

SECONDARY OUTCOMES:
significant improvement in writing | up to 1 week
  improvement of other quantitative test scores of writing (VAS subjective discomfort writing, DPRE scales and parameters measured on touchpad) after a single session of 1 Hz rTMS inhibitory to the left CSS , compared to the scores achieved in the 24 hours before the session of rTMS.
  Active or sham stimulation will be randomly assigned to the patient and the other session will be performed 3 days later.
improvement of dystonia on the scale WDRS | up to 1 week
  Assessing the improvement of dystonia on the scale WDRS after a single session of 1 Hz rTMS inhibitory to the left CSS, compared to the scores achieved in the 24 hours before the session of rTMS.
  Active or sham stimulation will be randomly assigned to the patient and the other session will be performed 3 days later.
correlation between the scores and the other parameters of disease severity | up to 1 week
  Assess whether age, disease duration and the presence of cortical atrophy are inversely correlated with the evolution of scores.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie KUBIS, MD, PhD, Study Director — Physiology Department, Lariboisière Hospital; Jean-Marc TROCELLO, MD, Principal Investigator — Neurology, Lariboisière Hospital
Locations (1):
- Hospital Lariboisiere, Paris, Île-de-France Region, France